CLINICAL TRIAL: NCT02417272
Title: Comparison of 2 Surgical Approaches in the Treatment of Cervical Degenerative Disc Disease: Total Disc Replacement Versus Anterior Cervical Decompression and Fusion
Brief Title: Total Disc Replacement Versus Anterior Cervical Decompression and Fusion
Acronym: CERVIDISC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2010/40
Record Dates: First submitted 2015-01-28; First posted 2015-04-15 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: Total Disc Replacement; Anterior Cervical Decompression and Fusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total disc replacement (TDR) (Experimental): Total disc replacement with preserved segmental motion decreasing load on adjacent levels.
  Interventions: Device: Surgical treatment of cervical degenerative disc disease (CP ESP®)
- Anterior Cervical Decompression and Fusion (ACDF) (Experimental): Interbody fusion by replacing disc space with a cage packed with bone substitute, and inserted into the anterior portion of the interspace.
  Interventions: Device: Surgical treatment of cervical degenerative disc disease (Axelle®)

INTERVENTIONS:
Device: Surgical treatment of cervical degenerative disc disease (CP ESP®)
  Arms: Total disc replacement (TDR)
Device: Surgical treatment of cervical degenerative disc disease (Axelle®) — Axelle®
  Arms: Anterior Cervical Decompression and Fusion (ACDF)

SUMMARY:
Background : Cervical degenerative disc disease is frequent and the consequence of aging. Degeneration may lead to disc herniation. Surgery is indicated in the presence of root compression with cervicobrachial neuralgia and/or myelopathy.

Purpose: The main objective of the study is the comparison of efficacy between total disc replacement (TDR) and Anterior Cervical Decompression and Fusion (ACDF) as surgical treatment of symptomatic cervical degenerative disc disease in term of "Success" rate, defined as preservation of adjacent segments, 24 months after surgery.

In our knowledge, there are no published data about randomized clinical trials comparing these radiological parameters (worsening of degeneration signs on static cervical spine radiographs and worsening of disc degeneration signs on MRI) at levels adjacent to surgery, between these 2 surgical approaches in patients suffering from cervical degenerative disc disease.

DETAILED DESCRIPTION:
Surgical treatment of cervical degenerative disc disease usually consists in neural decompression followed by intervertebral space reconstruction.

ACDF consists in interbody fusion by replacing disc space with a cage packed with bone substitute, and inserted into the anterior portion of the interspace. Fusion is successful in approximately 95% of patients with good to excellent clinical results in most of them. Unfortunately, up to 25% of these patients will develop degenerative changes at adjacent levels after surgery.

TDR consists in total disc replacement with preserved segmental motion decreasing load on adjacent levels.

Worsening of radiological degeneration signs at adjacent levels seems to be an important long term prognostic factor for reoperation.

In this trial, included patients will be randomly assigned to undergo either TDR or ACDF Six visits are planned during the study: pre inclusion visit within 3 months before surgery, inclusion/randomisation the day before surgery, 3 follow up visits (45 days, 6, and 12 months after surgery) and an end of study visit 24 months after surgery (or at time of withdrawal if relevant).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* suffering from cervical disc degenerative disease (whatever the grade, level and intervertebral disc height) needing one-level surgical treatment due to either invalidating cervicobrachial nevralgia despite 3-month optimal medical treatment or neurological symptoms, with motion of surgical level at least equal to 2° degrees, and non-degenerative adjacent discs.
* Being affiliated to health insurance
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)

Exclusion Criteria:

* Previous cervical traumatism and/or cervical surgery.
* Cervical degeneration defined as a Grade 4 according to modified Mehren classification and/or a Grade 5 according to Miyazaki et al classification on T2 magnetic resonance imaging (MRI), at symptomatic level and/or its adjacent levels.
* Myelopathy.
* Cervical spine instability.
* Presence of at least one major contraindication to surgery and/or general anaesthesia (ie, non-controlled coagulopathy, active infection, or serious underlying disease, auto-immune affection).
* Presence of at least one contraindication to either TDR or ACDF procedure.
* Presence of at least one contraindication to either static/dynamic radiographs or Magnetic Resonance Imaging (MRI).
* Severe radiological osteoporosis.
* Bone metabolic disease.
* Active cancer at time of inclusion into the study.
* Chronic intake of corticosteroids or any other treatment susceptible to interfere with study conduct and/or assessment (ie, immunosuppressive drugs).
* Unlikely to comply with the requirements of the study and/or to complete the study for psychological, social, familial or geographical reasons.
* No contraception for women of childbearing age
* Pregnant or breastfeeding women
* Being under guardianship or legal supervision.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
To compare efficacy of TDR and ACDF as surgical treatment of cervical degenerative disc disease in term of "success rate" defined as absence of radiological degenerative disease at adjacent levels | 24 months after surgery

SECONDARY OUTCOMES:
Between-group comparison of tolerance | 24 months after surgery
  This measure is a composite with :
  * Per- and post-operative surgery parameters
  * Major complication rate
  * Minor complication rate
Between-group comparison of efficacy | 45 days, 6, 12 and 24 months after surgery
  This measure is a composite with :
  * Cervical and radicular pain outcome as compared to preoperative status.
  * Functional outcome: Neck Disability Index (NDI) and modified Prolo Economic and Functional scores as compared to preoperative status.
  * Cervical radiological parameters
  * Quality of life outcome as compared to preoperative status.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine BENARD, MD, Study Chair — University Hospital Bordeaux, France; Olivier GILLE, Prof, Principal Investigator — University Hospital Bordeaux, France
Locations (3):
- France (3):
  - Chirurgie Orthopedique, Bordeaux
  - CHU Nice - Unité de Chirurgie Rachidienne, Nice
  - Chirurgie Orthopedique, Paris